CLINICAL TRIAL: NCT02593175
Title: Women's Triple-Negative First-Line Study: A Phase II Trial of Panitumumab, Carboplatin and Paclitaxel (PaCT) in Patients With Localized Triple-Negative Breast Cancer (TNBC) With Tumors Predicted Insensitive to Standard Neoadjuvant Chemotherapy
Brief Title: Women's MoonShot: Neoadjuvant Treatment With PaCT for Patients With Locally Advanced TNBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0294; NCI-2015-02183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0294 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (panitumumab, paclitaxel, carboplatin) (Experimental): Patients receive panitumumab IV over 30 minutes and paclitaxel IV over 30 minutes on days 1, 8, and 15. Patients also receive carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Biological: Panitumumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix

SUMMARY:
This phase II trial studies how well panitumumab, carboplatin and paclitaxel work in treating patients with newly diagnosed triple negative breast cancer that is limited to the breast and possibly to the nearby lymph nodes (locally advanced). This treatment study is linked to NCI-2015-00191 protocol, which uses a baseline biopsy to determine the neoadjuvant therapy that matches the sub-type of triple negative breast cancer (TNBC). Immunotherapy with panitumumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving panitumumab, carboplatin and paclitaxel before surgery may be an effective treatment for breast cancer by making the tumor smaller and reducing the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the pathologic complete response (pCR), residual cancer burden (RCB)-0 and RCB-I rates of patients with localized TNBC who were treated with panitumumab, carboplatin and paclitaxel (PaCT) in the neoadjuvant setting.

SECONDARY OBJECTIVES:

I. To estimate progression free survival (PFS) distribution of localized TNBC patients who were non-responders to initial anthracycline and cyclophosphamide chemotherapy, and who were treated with the PaCT regimen in the neoadjuvant setting.

II. Determine changes of epidermal growth factor receptor (EGFR) downstream biomarkers one week after 1 dose of panitumumab.

III. Determine response rate after 4 cycles of PaCT using radiographic imaging. IV. Correlate pathologic response with EGFR expression as measured by immunohistochemistry (IHC).

V. Determine toxicity associated to 4 cycles of PaCT in the neoadjuvant setting.

VI. Compare pathologic response to 4 cycles of PaCT in EGFR overexpressing tumors versus (vs.) non-EGFR overexpressing tumors.

VII. Compare pathologic response in tumors to 4 cycles of PaCT vs. 12 weeks of weekly paclitaxel (using data collected in conjunction with protocol 2014-0185).

EXPLORATORY OBJECTIVES:

I. Determine the correlation between EGFR expression by IHC and the presence of enhanced EGFR gene signatures at the time of initial tumor biopsy prior to neoadjuvant setting (NACT) (using gene expression data obtained from the protocol 2014-0185).

II. Determine rates of pCR in patients with EGFR overexpressed tumors identified by gene signatures (using gene expression data obtained from protocol 2014-0185) and compare to pCR rates in non-EGFR overexpressed tumors.

III. Determine the correlation between EGFR expression by IHC and the changes of EGFR downstream changes induced in surgery sample after completion of PaCT regimen.

IV. Determine the change in programmed cell death ligand 1 (PD-L1) glycosylation induced by panitumumab, and correlation with efficacy.

V. Determine the change after treatment in blood-based markers, if any, and use these to predict a response to panitumumab treatment.

OUTLINE:

Patients receive panitumumab intravenously (IV) over 30 minutes and paclitaxel IV over 30 minutes on days 1, 8, and 15. Patients also receive carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an intact evaluable primary tumor or biopsy proven axillary node involvement with at least 1.0 centimeter (cm) smallest dimension based on imaging after neoadjuvant anthracycline-based chemotherapy and prior to initiation of neoadjuvant chemotherapy under this protocol; baseline measurements and evaluations must be obtained within 4 weeks of registration to the study; all areas of disease should be recorded in order to assess response and uniformity of response to therapy
* Triple-negative breast cancer defined as estrogen receptor (ER) < 10%; progesterone receptor (PR) < 10% by immunohistochemistry (IHC) and human epidermal growth factor receptor 2 (HER2) 0-1 positive (+) by IHC or 2+, fluorescence in situ hybridization (FISH) < 2, gene copy number < 4
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have received at least one dose of an anthracycline based neoadjuvant regimen; patients are eligible if therapy was discontinued due to disease progression or therapy intolerance
* Baseline multi-gated acquisition (MUGA) or echocardiogram showing left ventricular ejection fraction (LVEF) >= 50% within 6 weeks prior to initiation of neoadjuvant chemotherapy
* Serum creatinine =< 1.5 mg/dl
* Creatinine clearance (CrCl) >= 50 mL/min calculated by the Cockcroft-Gault method
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 3.0 x upper limit of normal
* Alkaline phosphatase (Alp) =< 2.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Signed informed consent

Exclusion Criteria:

* Patient is unwilling or unable to sign and date the Institutional Review Board (IRB) approved informed consent
* Patients with less than a 1.0 cm measurable residual disease after neoadjuvant anthracycline based chemotherapy
* Women that are pregnant or lactating
* Patients with a history of prior malignancy within 5 years of study entry with the exception of curatively treated non-melanomatous skin cancer or carcinoma in situ of the cervix or breast
* Patients with a history of stage IV or metastatic disease
* Any serious medical illness, other than that treated by this study, which would limit survival to less than 1 month or psychiatric illness which would limit informed consent
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection
* Patients with a peripheral neuropathy > grade 1
* Patients with a history of serious cardiac events defined as: New York Heart Association class 3 or 4 heart failure, or history of myocardial infarction, unstable angina or cerebrovascular accident (CVA) within 6 months of protocol registration
* Patients with a history of PR prolongation or atrioventricular (AV) block
* Patients with a history of prior therapy with paclitaxel and/or carboplatin
* Patients who have received a cumulative dose of doxorubicin of greater than 360 mg/m^2 or epirubicin of greater than 640 mg/m^2
* Patients who concurrently use hormonal therapy and/or concurrent radiation therapy
* Patients who had prior radiation therapy of the primary breast carcinoma or axillary lymph nodes
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after; highly effective contraception methods include combination of any two of the following: placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository, total abstinence or male/female sterilization; women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to treatment; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Negative serum or urine pregnancy test for women within 72 hours of receiving the first dose of the study medication for women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yam C, Patel M, Hill HA, Sun R, Bassett RL Jr, Kong E, Damodaran S, Koenig KB, Abouharb S, Saleem S, Bisen AK, Murthy RK, Ramirez DL, Rauch GM, Adrada BE, Candelaria RP, Wang X, Mittendorf EA, Thompson AM, White JB, Ravenberg EE, Clayborn AR, Ding QQ, Booser DJ, Oke O, Brewster AM, Hortobagyi GN, Ibrahim NK, Litton JK, Valero V, Arun BK, Tripathy D, Chang JT, Chen K, Korkut A, Moulder SL, Huo L, Lim B, Ueno NT. Targeting the Epidermal Growth Factor Receptor Pathway in Chemotherapy-Resistant Triple-Negative Breast Cancer: A Phase II Study. Cancer Res Commun. 2024 Oct 1;4(10):2823-2834. doi: 10.1158/2767-9764.CRC-24-0255. PMID 39356138
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment took place in the Breast Medical Oncology clinics of MD Anderson Cancer Center locations from November of 2016 through August of 2021
Groups:
- Panitumumab Plus Carboplatin and Paclitaxel: Patients receive panitumumab 2.5mg/kg IV and paclitaxel 80mg/kg IV weekly x 12 weeks, and carboplatin AUC4 IV q3w x 4 cycles
Period: Overall Study
Arm/Group | Panitumumab Plus Carboplatin and Paclitaxel
Started | 43
Completed | 34
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Disease progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 48.6 [26 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 25
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Residual Disease
Description: Residual Disease at the time of surgery, which can help predict disease recurrence and survival across all breast cancer subtypes.
Time Frame: At the time of surgery
Population: All patients were evaluable for data analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab Plus Carboplatin and Paclitaxel
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Panitumumab Plus Carboplatin and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 2/43
Other Adverse Events (participants affected / at risk) | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab Plus Carboplatin and Paclitaxel (N=43)
Cystitis (Renal and urinary disorders) | 1 (2)
Vertigo (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab Plus Carboplatin and Paclitaxel (N=43)
Neutrophil Count decreased (Investigations) | 22 (31)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (21)
Fatigue (General disorders) | 22 (22)
Anemia (Blood and lymphatic system disorders) | 17 (26)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 20 (20)
Mucositis Oral (Gastrointestinal disorders) | 27 (27)
Dry Skin (Skin and subcutaneous tissue disorders) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT02593175/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT02593175/ICF_000.pdf